CLINICAL TRIAL: NCT05773196
Title: SAN-09611: Prospective Single-Timepoint Huntington's Disease Biospecimen Collection Study
Brief Title: Prospective Single-Timepoint Huntington's Disease Biospecimen Collection Study
Acronym: SAN-09611
Status: Recruiting | Type: Observational
Sponsor: Sanguine Biosciences (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-09611
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Huntington Disease; Huntington's Dementia; Huntington Disease, Late Onset; Huntington; Dementia (Etiology)
MeSH Terms: conditions — Huntington Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cohort 1-Huntington's Disease:
  The target blood volume of each phlebotomy visit will be 20 mL. The minimum accepted volume (in the event of tough venipuncture attempts or difficulty obtaining the blood) will be 5 mL. The maximum amount that can be drawn in a 6-week period will be 100 mL (whole blood 6-week maximum).
  Sample Collection:
  * 10 mL EDTA Vial (Box 1; Frozen)
    o Whole blood will be collected into 1 x 10 ml EDTA tube (no in-home/laboratory processing), shipped frozen (on dry ice) FedEx priority overnight (by 10:30 am) to Labcorp after each collection in box 1.
  * 10 mL EDTA Vial (Box 2; Ambient)
    * Whole blood will be collected into 1 x 10 ml EDTA tube (no in-home/laboratory processing), shipped ambient FedEx priority overnight (by 10:30 am) to Labcorp after each collection in box 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biospecimen Collection — Cohort 1-Huntington's Disease:
  The target blood volume of each phlebotomy visit will be 20 mL. The minimum accepted volume (in the event of tough venipuncture attempts or difficulty obtaining the blood) will be 5 mL. The maximum amount that can be drawn in a 6-week period will be 100 mL (whole blood 6-week maximum).
  Sample Collection:
  * 10 mL EDTA Vial (Box 1; Frozen)
    o Whole blood will be collected into 1 x 10 ml EDTA tube (no in-home/laboratory processing), shipped frozen (on dry ice) FedEx priority overnight (by 10:30 am) to Labcorp after each collection in box 1.
  * 10 mL EDTA Vial (Box 2; Ambient)
    * Whole blood will be collected into 1 x 10 ml EDTA tube (no in-home/laboratory processing), shipped ambient FedEx priority overnight (by 10:30 am) to Labcorp after each collection in box 2.

SUMMARY:
OBJECTIVES:

The primary study objective is to collect blood from participants with Huntington's Disease in order to validate a CE marked Cytosine, Adenine, Guanine (CAG) assay for use in future studies for Huntington's Disease.

The secondary study objective is to create a biorepository that can be used to identify disease associated biomarkers and potential targets with immune and multi-omics profiling. The disease sample collection and analysis will be the foundation for an extensive network of biospecimen access and linked datasets for future translational research.

DETAILED DESCRIPTION:
STUDY DESIGN:

* This protocol is a single-center, single-cohort, bioresearch study enrolling up to 5 participants. The cohort is as follows:

  o Cohort 1: Huntington's Disease (n=5)
* The study will enroll participants per the eligibility criteria.
* Participants will have 1 scheduled biospecimen collection visit(s). If the participant requires a recollection or is called for an extra sample donation, this will add additional volume and visit(s) to the collection schedule. The biospecimens collected from participants are whole blood.
* The target blood volume of each phlebotomy visit will be 20 mL. The minimum accepted volume (in the event of tough venipuncture attempts or difficulty obtaining the blood) will be 5 mL. The maximum amount that can be drawn in a 6-week period will be 100 mL (whole blood 6-week maximum).
* Confirmation of eligibility and medical record review by a member of the study staff will be completed for participants of the cohort before they are considered fully enrolled.

ELIGIBILITY:
Cohort 1: Huntington's Disease

Inclusion:

1. The participant is willing and able to provide written informed consent
2. The participant is willing and able to provide appropriate photo identification
3. Participants aged 25 to 65, inclusive
4. Participants have been diagnosed with Huntington's Disease
5. Patients must have numerical documentation of CAG repeats present in the Medical Record, along with a Huntington's Disease diagnosis.
6. Pre-existing evidence of CAG repeats should be in the range of 40-60 repeats *Preference (not required for enrollment): Patients to have different CAG repeats from each other but this is not essential.*

Exclusion:

1. Participants who are pregnant or are nursing
2. Participants with a known history of HIV, hepatitis, or other infectious diseases
3. Participants who have taken an investigational product in the last 30 days
4. Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The biospecimen subtypes for this study include whole blood from people diagnosed with Huntington's disease. The global prevalence and rising burden of Huntington's disease is a worldwide healthcare concern. Huntington's Disease is seen as frequently in 10.6-13.7 people per 100,000 individuals.10 The collection and analysis of samples from the diseased specimens will lay the groundwork for an extensive network of biospecimen access and linked datasets for future translation research in therapeutic development and a better understanding of the disease to improve health outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Biospecimen Collection | 6 months
  The primary study objective is to collect blood from participants with Huntington's Disease in order to validate a CE marked Cytosine, Adenine, Guanine (CAG) assay for use in future studies for Huntington's Disease.

SECONDARY OUTCOMES:
Biorepository creation | 6 months
  The secondary study objective is to create a biorepository that can be used to identify disease associated biomarkers and potential targets with immune and multi-omics profiling. The disease sample collection and analysis will be the foundation for an extensive network of biospecimen access and linked datasets for future translational research.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanguine Biosciences, Inc., Woburn, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data provided to Roche only.